CLINICAL TRIAL: NCT04767906
Title: Cabozantinib Treatment in a Phase II Study for Patients With Hepatocellular Carcinoma (HCC) Refractory to PD-1 Inhibitors
Acronym: CaPture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaPture
Record Dates: First submitted 2021-01-08; First posted 2021-02-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC, Cabozantinib, PD-1 inhibitor, PD-L1 inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Patients with hepatocellular carcinoma with prior non-response or disease progression during a PD-1 or PD-L1 inhibitor treatment will be treated with Cabozantinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Other): Enrolled patients start with 60mg of Cabozantinib. The maximum duration of treatment is 336 days. The dose can be adjusted by the physician to 40mg or 20mg.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — The medication is taken once a day for 336 days (max.). The start dose is 60mg and can be reduced according to the physicians decision. 40mg and 20mg are also available.

SUMMARY:
The CaPture trial is a prospective, multi-centre, non-randomized phase II study. Its aim is to assess feasibility, safety and efficacy signals of Cabozantinib treatment in patients with HCC and prior non-response or disease progression during a PD-1 or PD-L1 inhibitor treatment. Since the potential study population is very small, the sample size has been fixed in advance to N = 40. Time on treatment (TT) will be measured as primary endpoint.

DETAILED DESCRIPTION:
Patients will be recruited at the participating trial sites (up to ten trial sites), which are all specialized in treatment of patients with HCC. Once potential patients are identified by trial physicians, they will be asked for trial participation and informed consent by one investigator of the CaPture trial. Patients included within 4 weeks after diagnosis of failure of preceding PD-1/PD-L1 inhibitory treatment.

After baseline, visits are previewed on a 4weekly (28 days) basis during the whole duration of Cabozantinib study treatment, which can be used for a maximum of 12 months (336 days). The treatment with Cabozantinib will be performed in accordance with the valid license and according to the judgement of the treating physician.The tablet is taken once a day, starting normally with the highest dosage (60 mg). The doses 20mg and 40mg are still available and can be used for dose reduction. During the visits, the patient will be questioned for compliance and side effects and examined for clinical and laboratory parameters.

Response to Cabozantinib should be assessed at least every 12 weeks (84 days) by either CT scan or MRI.

After termination of Cabozantinib study treatment the first follow-up visit takes place one month after the end of therapy in person. Further follow-up visits can be done by phone to collect patient's status and further treatment.

In addition to the time on treatment (TT), survival, response, feasibility, biomarkers, health status and safety should also be tested.

Furthermore there is an concomitant scientific project. The aim of this project is to examinate the association of HCC related biomarkers with response to Cabozantinib in patients treated in the CaPture study. For this, we will analyse liver biopsy samples as well as circulating markers in patients who are willing to participate in the project.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of locally advanced or metastatic and/or unresectable hepatocellular carcinoma (HCC)
2. Pre-Treatment with a PD-1/PD-L1 inhibitor for at least one administration which was given as first line or as following line systemic treatment alone or in combination with other systemic or local treatments (e.g. TACE)
3. Disease progression or end of therapy due to toxicity during/after pre-therapy
4. CTCAE ≤ Grade 2 prior to study registration, with the exception of alopecia
5. ECOG (Eastern Cooperative of Onco-logy Group) Index 0 or 1
6. Age ≥ 18 years
7. Written informed consent

Exclusion Criteria:

1. Significant portal hypertension (moderate or severe ascites)
2. No adequate controlled arterial hypertension (RR > 140/80mmHg)
3. ALAT/ASAT five times higher then upper normal value
4. Hepatic encephalopathy (every stage)
5. Liver cirrhosis Child-Pugh B and C
6. Known fibrolamellar HCC, sarcomatoid HCC, or cholangiocarcinoma mixed with HCC
7. Major surgical procedure, other than for diagnosis, within eight weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
8. Severe infection with alteration of general condition within four weeks prior to initiation of study treatment
9. Severely impaired kidney function (CDK: stadium 4: GFR<30)
10. Myocardial infarction within 12 months prior to initiation of study treatment
11. Epilepsy
12. Heart failure, Cardiac arrhythmia, respectively long-QT syndrome
13. Severe bleeding or high risk for the development of severe bleeding, including esophageal varices > 1° or esophageal varices with red marks as seen on a lighted stomach scope (endoscopy)
14. Chronic inflammatory bowel disease (e.g. colitis ulcerosa, diverticulitis, Crohn's disease)
15. Increased risk of thromboembolism due to medical history or disease
16. Significant alcohol consumption (>1 drink/day; 1 drink=0.25l beer or 0,1l wine or 2cl spirituous beverages)
17. Known active HIV infection
18. Known hereditary galactose intolerance, lactase deficiency, glucose-galactose malabsorption
19. Prior Cabozantinib use
20. Ongoing therapy with direct oral anticoagulants (DOAK) / platelet aggregation inhibitor or statine (e.g. Ticagrelor, Clopidogrel)
21. Predicted life expectancy of less than 6 months
22. Female patients who do not meet at least one of the following criteria:

    * Postmenopausal women (for at least 1 year before the screening visit) OR
    * Postoperative status (6 weeks after bilateral ovariectomy with or without hysterectomy) OR
    * If they are of childbearing potential, agree to practice one highly effective method of contraception and one additional effective (barrier) method at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.) OR
    * Abstinence OR
    * Vasectomy of the partner
23. Male patients not using one of the following variants for contraception including a period of 4 months after the completion of the therapy:

    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. OR
    * Condition after vasectomy OR
    * Condom
24. Participation in any other interventional trials within 28 days prior to initiation of study treatment
25. Suspected lack of compliance to previous treatments; inability to take the medication
26. Pregnancy or lactation, or intention of becoming pregnant during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
time on treatment (TT) | start of treatment until end of treatment (max. 336 days)
  Primary endpoint of the trial is the time on treatment (TT). TT is defined as one plus the last date of treatment with Cabozantinib minus the first date of treatment with Cabozantinib, and will be measured in days (note that Cabozantinib will be administered as a single dose per day). The end of treatment must be confirmed by the investigator. In particular, planned discontinuations or missing compliance will not be considered as end of treatment without confirmation.

SECONDARY OUTCOMES:
Overall survival (OS) | screening visit until date of death, maximum until the last registered patient reached the second follow-up (6 months after end of therapy)
  Overall survival (OS), is the time to death of any cause. OS is measured in days, defined as death date minus registration date.
Progression-free survival (PFS) | screening visit until the time to tumor progression or date of death from any cause, whichever came first, maximum until the last registered patient reached the second follow-up (6 months after end of therapy)
  Progression-free survival (PFS) is the time to tumor progression or death of any cause, whichever comes first. PFS is measured in days, defined as date of diagnosis of tumor progression by mRECIST criteria minus registration date. If a patient dies without previous diagnosis of tumor progression, date of diagnosis is replaced by death date.
Duration of response (DoR) | screening visit until the time from achievement of response or date of death from any cause, whichever came first, maximum until the last registered patient reached the second follow-up (6 months after end of therapy)
  is the time from achievement of response (i.e., measurement criteria for CR or PR are first met, cf. Eisenhauer et al., 2009, p. 236) until the first date that tumor recurrence or progression is documented (taking as reference the smallest measurements recorded in the study) or death of any cause, whichever comes first. DoR is measured in days, defined as date of documentation of tumor progression by mRECIST criteria minus date of documentation of tumor response (CR or PR). If a patient dies without previous diagnosis of tumor progression, date of progression documentation is to be replaced by death date. If CR or PR will never be documented for a patient, DoR is set to "zero".
Response rates | screening visit until end of treatment (max. 336 days)
  Response rates, measured in percent, are defined as the number of patients whose best tumor response observed by mRECIST criteria is CR, PR, SD or PD, respectively, divided by the total number of registered patients. The overall response rate (ORR) is defined as the number of patients whose best tumor response observed by mRECIST criteria is CR or PR divided by the total number of registered patients.
Median average dose | start of treatment until end of treatment (max. 336 days)
  Median average dose, measured in milligram (mg). Averages of all Cabozantinib doses administered will be calculated weekly from first date of treatment until end of treatment. Discontinuations of treatment for any reason, including missing compliance, will be included into this calculation as zero doses. Median average dose is defined as the median of the obtained sequence of averages.
Image-based endpoint: Tumor progression | screening until end of treatment (max. 336 days)
  Tumor progression, assessed at Visits 3, 6, 9, 12 and EoT visit (if applicable) in comparison to the state at Screening, by mRECIST criteria.
Image-based endpoint: Progression of tumoral macrovascular invasion | screening until end of treatment (max. 336 days)
  Progression of tumoral macrovascular invasion of hepatic and/or portal vein branches, assessed at Visits 3, 6, 9, 12 and EoT visit (if applicable) according to the working instruction for radiologists, in comparison to state at Screening.
Image-based endpoint: Progression of extrahepatic HCC manifestations | screening until end of treatment (max. 336 days)
  Progression of extrahepatic HCC manifestations, assessed at Visits 3, 6, 9, 12 and EoT visit (if applicable) according to the working instruction for radiologists, in comparison to state at Screening.
Image-based endpoint: Total tumor volume | screening until end of treatment (max. 336 days)
  Total tumor volume (TTV), assessed at Screening, Visits 3, 6, 9, 12 and EoT visit (if applicable), measured in cm^3 according to the working instruction for radiologists.
Image-based endpoint: Affection rate | screening until end of treatment (max. 336 days)
  Affection rate, assessed at Screening, Visits 3, 6, 9, 12 and EoT visit (if applicable), measured in percent. Affection rate is defined as total tumor volume divided by total liver volume, both measured in cm^3 according to the working instruction for radiologists.
Concentration of Alpha-fetoprotein (AFP), | screening until end of treatment (max. 336 days)
  Concentration of Alpha-fetoprotein (AFP), measured in µg/l, at Screening and Visits 0, 3, 6, 9, 12 and EoT visit (if applicable).
Child-Pugh classification score | screening until first follow-up (one month after EoT)
  Child-Pugh classification score, measured in levels from A to C, at Screening and Visits 3, 6, 9, 12, EoT and FU1 (if applicable).
ECOG Performance Status | screening until first follow-up (one month after EoT)
  ECOG Performance Status, measured in levels from 0 to 5, at Screening and Visits 3, 6, 9, 12, EoT and FU1 (if applicable).
drug-related interruption, reduction or termination of treatment (safety endpoint) | start of treatment until end of treatment (max. 336 days)
  Descriptive documentation
occurence of clinical symptoms of liver dysfunction (safety endpoint) | start of treatment until end of treatment (max. 336 days)
  Descriptive documentation

CONTACTS AND LOCATIONS:
Overall Officials: Florian van Bömmel, MD, Study Chair — Authorised representative of the sponsor (University of Leipzig)
Locations (5):
- Germany (5):
  - Technische Universität Dresden, Medizinische Fakultät Carl Gustav Carus Medizinische Klinik und Poliklinik I, Dresden, Saxony
  - MVZ Mitte/MVZ Delitzsch GmbH, Leipzig, Saxony
  - University Hospital Leipzig, Leipzig, Saxony
  - Charite Universitätsmedizin, Campus Virchow Klinikum, Klinik für Hepatologie/Gastroenterologie, Berlin
  - Universitätsklinikum Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: Yes
After publication of the major results and upon reasonable request from researchers performing an individual patient data meta-analysis, individual patient data underlying published results will be shared after re-identification. This requires approval by the local Institutional Review Board (IRB) of the researcher requesting the data along with public registration of the meta-analysis.
Supporting Information: Study Protocol, CSR
Time Frame: After publication of the major results.
Access Criteria: Individual patient data underlying published results will be shared after re-identification. This requires approval by the local Institutional Review Board (IRB) of the researcher requesting the data along with public registration of the meta-analysis.